CLINICAL TRIAL: NCT05262062
Title: Effect of Integrated Neuromuscular Inhibition, Muscle Energy and Strain Counter Strain Techniques in the Management of Mechanical Neck Pain.
Brief Title: Integrated Neuromuscular Inhibition, Muscle Energy and Strain Counter Strain Techniques in Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Zainab Mahmood
Record Dates: First submitted 2022-02-20; First posted 2022-03-02 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Neck Pain
Keywords: Mechanical Neck Pain; Chronic Neck Pain; Muscle Energy Technique; Strain counter Strain; INIT
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Strain Counter Strain Technique (Experimental): When general or local pain began to diminish, upper trapezius , levator scapulae and SCM was placed in a position of ease and was held for approximately 20 to 30 seconds.
  Moderate digital pressure was applied to the identified MTrP as participants rated their level of pain on a scale ranging from 1 to 10.3. Ease was defined as the point at which a reduction in pain of at least 70% was achieved.Once the position of ease was identified, it was held for 20 to 30 seconds.
  Interventions: Other: Strain Counter Strain Technique
- Muscle Energy Technique, (Experimental): After the ease position was maintained for 20 to 30sec an isometric contraction focused on the muscle fibers around the MTrP was performed.
  Each isometric contraction was held for 7 to 10 sec and was followed by a soft-tissue stretch for 15 seconds and then relax for 30 seconds. Each stretch was held for 30 seconds, and it was repeated 3 times during the treatment session.
  3. Treatment was performed on the 3 most painful areas between the upper border of the upper trapezius muscle, the SCM, the levator scapulae, and the SC muscle.
  Interventions: Other: Muscle Energy Technique,
- Integrated Neuromuscular Inhibition Technique (Experimental): 1. Group c will receive Combination of exercise (strain counter strain , muscle energy & ischemic compression. In ischemic compression patient will receive compression,2. After MTrPs identification, 3. Ischemic compression was applied in an intermittent manner for up to 2 minutes for each MTrP.
  4. The pincer grasp (for the trapezius muscle and SCM) or direct digital pressure (for the levator scapulae and SC muscle) was used with the patients in either the supine position or sitting upright.
  Interventions: Other: Integrated Neuromuscular Inhibition Technique

INTERVENTIONS:
Other: Strain Counter Strain Technique — When general or local pain began to diminish, upper trapezius , levator scapulae and SCM was placed in a position of ease and was held for approximately 20 to 30 seconds.
  2. Moderate digital pressure was applied to the identified MTrP as participants rated their level of pain on a scale ranging from 1 to 10.
  3. Ease was defined as the point at which a reduction in pain of at least 70% was achieved.
  4. Once the position of ease was identified, it was held for 20 to 30 seconds.
  Arms: Strain Counter Strain Technique
Other: Muscle Energy Technique, — After the ease position was maintained for 20 to 30sec an isometric contraction focused on the muscle fibers around the MTrP was performed.
  2. Each isometric contraction was held for 7 to 10 sec and was followed by a soft-tissue stretch for 15 seconds and then relax for 30 seconds. Each stretch was held for 30 seconds, and it was repeated 3 times during the treatment session.
  3. Treatment was performed on the 3 most painful areas between the upper border of the upper trapezius muscle, the SCM, the levator scapulae, and the SC muscle.
  Arms: Muscle Energy Technique,
Other: Integrated Neuromuscular Inhibition Technique — 1. Group c will receive Combination of exercise (strain counter strain , muscle energy & ischemic compression. In ischemic compression patient will receive compression,
  2. After MTrPs identification,
  3. Ischemic compression was applied in an intermittent manner for up to 2 minutes for each MTrP.
  4. The pincer grasp (for the trapezius muscle and SCM) or direct digital pressure (for the levator scapulae and SC muscle) was used with the patients in either the supine position or sitting upright
  Arms: Integrated Neuromuscular Inhibition Technique

SUMMARY:
1. To determine effects of Neuromuscular Inhibition, Muscle energy and strain counter strain techniques on Pain, disability, pain pressure threshold, range of motion, and health-related quality of life in mechanical neck pain.
2. To compare the effects of Integrated Neuromuscular inhibition, Muscle energy and strain counter strain techniques in the Management of mechanical neck pain.

ELIGIBILITY:
Inclusion Criteria:

* Participants falling in this category would be recruited into the study.

  * Patients with chronic mechanical neck pain (symptoms for more than 3 months).
  * Age group between 30 - 60 years.
  * Patients willing to participate and take treatment.
  * Patients must have at least 1 active trigger point at upper trapezius, levator scapulae, SCM.
  * Gender (Both)
  * VAS >3

Exclusion Criteria:

* • Patients having severe neck pain.

  * Patients having any systemic joint pathology, inflammatory joint disease (e.g rheumatoid arthritis, gouty arthritis, psoriatic arthritis).
  * Patients who had any neurological deficit, myelopathy any mental illness.
  * Patients on medication like antidepressants, corticosteroid, anti-inflammatory medications.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2022-03-24 (Actual); Study Completion 2022-03-28 (Actual)

PRIMARY OUTCOMES:
• Visual analog scale. | 4 weeks
  Pain was assessed by the VAS, which is a card with an uncalibrated scale ranging from 0 to 10. 0 represent no pain and 10 represent the highest level of pain. A vertical line on the scale drawn by the patient marked their subjective pain estimation ranging from 0 to 10. Subsequently, a single ruler was used to record the exact pain level. The reliability of the scale is quite satisfactory, especially in people with moderate and high educational levels (r = .94, P = .001) (6). reference for tools should be added
• Neck disability index. | 4 Weeks
  Disability was evaluated using the NDI questionnaire. It is a self-reported 10-item scale. Each item assesses different neck pain complaints. Most of the items are related to restrictions in activities of daily life, and each item is expressed by 6 different assertions in the range 0 to 5, with 0 indicating no disability and 5 indicating the highest disability. The total score ranges from 0 to 50. Its credibility in people with neck pain is moderate to high and has been considered a valid tool in patients with neck problems. NDI has high reliability i.e. ICC 0.97 and good internal validity i.e. Cronbach's alpha = 0.86.(6)
• 36-Item Short Form Health Survey score | 4 Week
  SF-36 consists of 36 questions, selected from the Medical Outcomes Study. These questions are related to 8 different parameters of mental and physical health.SF-36 has satisfactory support in the literature.51 Total Physical and Mental Health, and the subcategory of Bodily Pain, were evaluated in this study. SF-36 shows a high rate of validity and reliability in patients with neck pain. In all 8 categories, both the ICC and the Cronbach's alpha index are high 0.75-0.94 and 0.69-0.88, correspondingly
• Goniometer | 4 Week
  Goniometer measures the available range of motion of cervical flexion, extension, rotation and side bending. To see the restriction in cervical moments we compare the available ROM's to the normal ROM's.
algometer | 4th Week
  Pressure pain threshold is measured by Pressure algometry was conducted using a Wagner digital algometer (Wagner FPX 25 Digital Algometer; Wagner Instruments, Greenwich, CT). PPT was assessed bilaterally over the upper border of the trapezius muscle, halfway between the midline and the lateral border of the acromion, the levator scapulae muscle 2 cm above the lower insertion and located in the upper medial border of the scapulae, the SCM upper insertion, and the SC 2 cm lateral to the spinous processes of the axis. The metal rod of the algometer was placed vertically on the site, and the examiner applied gradually increasing pressure at a rate of 1 kg/s. The examinees indicated when they began to feel pain or discomfort. Then, the examiner ceased the pressure and noted the value. Pressure algometry showed from satisfactory to fairly high reliability by various researchers both in repeated measurements of the same examiner and between measurements of different examiners.(14)

CONTACTS AND LOCATIONS:
Overall Officials: Lal Gul Khan, MSPT, Principal Investigator — Riphah International University Islamabad
Locations (1):
- Atta Memorial Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jahre H, Grotle M, Smedbraten K, Dunn KM, Oiestad BE. Risk factors for non-specific neck pain in young adults. A systematic review. BMC Musculoskelet Disord. 2020 Jun 9;21(1):366. doi: 10.1186/s12891-020-03379-y. PMID 32517732
- [Background] 2. Lin CC, Hua SH, Lin CL, Cheng CH, Liao JC, Lin CF. Impact of prolonged tablet computer usage with head forward and neck flexion posture on pain intensity, cervical joint position sense and balance control in mechanical neck pain subjects. Journal of Medical and Biological Engineering. 2020 Jun;40(3):372-82
- [Background] Aker PD, Gross AR, Goldsmith CH, Peloso P. Conservative management of mechanical neck pain: systematic overview and meta-analysis. BMJ. 1996 Nov 23;313(7068):1291-6. PMID 8942688
- [Background] Ashfaq R, Riaz H. Effect of Pressure biofeedback training on deep cervical flexors endurance in patients with mechanical neck pain: A randomized controlled trial. Pak J Med Sci. 2021 Mar-Apr;37(2):550-555. doi: 10.12669/pjms.37.2.2343. PMID 33679948
- [Background] Safiri S, Kolahi AA, Hoy D, Buchbinder R, Mansournia MA, Bettampadi D, Ashrafi-Asgarabad A, Almasi-Hashiani A, Smith E, Sepidarkish M, Cross M, Qorbani M, Moradi-Lakeh M, Woolf AD, March L, Collins G, Ferreira ML. Global, regional, and national burden of neck pain in the general population, 1990-2017: systematic analysis of the Global Burden of Disease Study 2017. BMJ. 2020 Mar 26;368:m791. doi: 10.1136/bmj.m791. PMID 32217608
- [Background] 6. Fryer G. Muscle energy technique: An evidence-informed approach. International Journal of Osteopathic Medicine. 2011 Mar 1;14(1):3-9.
- [Background] 7. Paul J, Balakrishnan P. Effect of strain counter strain technique and stretching in treatment of patients with upper trapezius tenderness in neck pain. INTERNATIONAL JOURNAL OF PHYSIOTHERAPY. 2018 Aug 1;5(4):141-4.
- [Background] 8. Ganjave P, Shikrapurkar S. Prevalence of Neck Pain among Clinical Laboratory Technicians in Mumbai
- [Background] Lytras DE, Sykaras EI, Christoulas KI, Myrogiannis IS, Kellis E. Effects of Exercise and an Integrated Neuromuscular Inhibition Technique Program in the Management of Chronic Mechanical Neck Pain: A Randomized Controlled Trial. J Manipulative Physiol Ther. 2020 Feb;43(2):100-113. doi: 10.1016/j.jmpt.2019.03.011. Epub 2020 May 30. PMID 32482433
- [Background] 10. Nugraha MH, Antari NK, Saraswati NL. The Efficacy Of Muscle Energy Technique In Individuals With Mechanical Neck Pain: A Systematic Review. Sport and Fitness Journal. 2020;8(2):91-8
- [Background] 11. Gohil D, Vaishy S, Baxi G, Samson A, Palekar T. Effectiveness of strain-counterstrain technique versus digital ischemic compression on myofascial trigger points. Archives of Medicine and Health Sciences. 2020 Jul 1;8(2):191.
- [Background] 12. Kumar GY, Sneha P, Sivajyothi N. Effectiveness of Muscle energy technique, Ischaemic compression and Strain counterstrain on Upper Trapezius Trigger Points: A comparative study. International journal of physical education, sports and Health. 2015;1(3):22-6.
- [Background] Toprak Celenay S, Mete O, Sari A, Ozer Kaya D. A comparison of kinesio taping and classical massage in addition to cervical stabilization exercise in patients with chronic neck pain. Complement Ther Clin Pract. 2021 May;43:101381. doi: 10.1016/j.ctcp.2021.101381. Epub 2021 Apr 2. PMID 33831805
- [Background] Nunes AMP, Moita JPAM, Espanha MMMR, Petersen KK, Arendt-Nielsen L. Pressure pain thresholds in office workers with chronic neck pain: A systematic review and meta-analysis. Pain Pract. 2021 Sep;21(7):799-814. doi: 10.1111/papr.13014. Epub 2021 May 6. PMID 33829681